CLINICAL TRIAL: NCT06896487
Title: THE EFFECT OF SUPERFICIAL EMG BIOFEEDBACK TRAINING ON MUSCLE ACTIVATION, PROPRIOCEPTION, REACTION TIME AND UPPER EXTREMITY FUNCTIONS IN PATIENTS WITH CHRONIC NECK PAIN: A SINGLE-BLIND RANDOMIZED CONTROLLED TRIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pervin Yeşiloğlu (Other)
Collaborators: Dokuz Eylul University (Other)
Responsible Party: Sponsor-Investigator, Pervin Yeşiloğlu, Research Assistant, Yuzuncu Yil University
Organization: Yuzuncu Yil University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: YYUPY01
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Chronic Neck Pain
MeSH Terms: interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Surface EMG Bofeedback Muscle and Relaxation Training (Experimental): Participants in this group were given muscle training and relaxation training for 6 weeks with superficial EMG Biofeedback protocol in addition to home exercise therapy.
  Interventions: Other: Surface EMG Biofeedback Muscle and Relaxation Training
- Conventional Rehabilitation Group (Experimental): Patients in this study group were enrolled in a conventional therapy program consisting of ultrasound, TENS and hot pack in addition to home exercise therapy.
  Interventions: Other: Conventional Rehabilitation
- Home Exercise Group (No Intervention): Patients in this group were only told about home exercises and asked to do them 3 days a week.

INTERVENTIONS:
Other: Surface EMG Biofeedback Muscle and Relaxation Training — We think that 6 weeks of superficial EMG Biofeedback muscle training and relaxation training given to the participants in this study will improve the patient's upper trapezius activation and voluntary contraction performance.
  Arms: Surface EMG Bofeedback Muscle and Relaxation Training
Other: Conventional Rehabilitation — The conventional rehabilitation group of this study received ultrasound, TENS and hot pack application 3 days a week for 6 weeks.
  Arms: Conventional Rehabilitation Group

SUMMARY:
Musculoskeletal disorders are among the health problems that most distract individuals from work life in both developed and developing countries. According to the 2019 Global Burden of Disease Study, when evaluated in terms of burden of disease, life expectancy with disability and rehabilitation needs, low back and neck pain are at the top of this category. According to the Health Research Report published by the Turkish Statistical Institute (TurkStat) in 2019, musculoskeletal disorders in the neck region are more common in women and were determined as the musculoskeletal disorder with the highest increase by 12.9% between 2016 and 2019.

It has been reported that in approximately half of individuals with neck pain, this pain recurs and becomes chronic. Factors such as sedentary lifestyle, history of low back pain, being female, anxiety disorders, sleep problems and smoking are thought to contribute to the chronicization of pain. Chronic neck pain is defined as pain in the neck region lasting longer than twelve weeks.

Cervical muscle activations have been monitored with EMG studies in the patient population with neck pain from past to present and altered cervical muscle activations have been reported in individuals with neck pain. The main muscle groups in which muscle activation has been monitored with superficial EMG and changes have been found in individuals with neck pain are upper trapezius, sternocelidomastoid, cervical erector spinal muscles and thoracic erector spinal muscles. On the other hand, it is still debated whether these muscle activation changes are the cause or a normal consequence of chronic neck pain.

In recent years, it has been reported in the literature that EMG Biofeedback studies have been included in patients with neck pain, but more studies are needed to determine its superiority to conventional applications. In the light of this information, in our study titled "The Effect of Superficial EMG Biofeedback Training on Muscle Activation, Proprioception, Reaction Time and Upper Extremity Functions in Patients with Chronic Neck Pain; Randomized controlled study", both the effect of EMG Biofeedback muscle training application on the symptoms of patients with neck pain will be investigated and data that will be a reference for future studies in this field will be obtained.

The study in patients with chronic neck pain had two aims. To investigate the effect of EMG Biofeedback relaxation training (upper trapezius muscle) combined with active EMG Biofeedback exercises + routine exercise program on muscle activation, pain, proprioception, reaction time and upper extremity function in patients with neck pain. To compare the effects of EMG Biofeedback training with standard physiotherapy program.

Hypotheses of the study; H0: EMG Biofeedback relaxation training (upper trapezius muscle) combined with active EMG Biofeedback exercises + routine exercise program has no effect on muscle activation, pain, proprioception, reaction time and upper extremity function in patients with neck pain H1: EMG Biofeedback relaxation training (upper trapezius muscle) combined with active EMG Biofeedback exercises + routine exercise program has an effect on muscle activation, pain, proprioception, reaction time and upper extremity function in patients with neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Presentation to the clinic with neck pain for at least 3 months due to at least one of the following causes: facet joint dysfunction, cervical disc lesions, myofascial pain syndrome, cervical spondylosis, mechanical neck pain,
* To be between the ages of 18-65,
* To cooperate with the evaluation parameters to be applied in the study,
* Volunteering to participate in the study,
* Not having received physical therapy for neck pain before,

Exclusion Criteria:

* Over 65 years of age,
* Problems in perceiving verbal commands,
* Having benefited from physiotherapy and/or another treatment method for neck pain within the last 1 year,
* Undergoing any operation related to pathologies of the neck region,
* To have undergone upper extremity surgery,
* Presence of neurological symptoms,
* Presence of comorbidities affecting upper extremity and hand functions (carpal tunnel syndrome, trigger finger, impingement syndrome, thoracic outlet syndrome, lateral and medial epicondylitis, hand osteoarthritis),
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-07-26 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Upper Extremity Reaction Time | Week of enrollment and end of the treatment at 6th weeks and 12 th weeks
Cervical Proprioception | Week of enrollment and end of the treatment at 6th weeks and 12 th weeks

SECONDARY OUTCOMES:
Range of Motion Assessment | Week of enrollment and end of the treatment at 6th weeks and 12 th weeks
Neck Pain and Disability Index | Week of enrollment and end of the treatment at 6th weeks and 12 th weeks
Neck Disability Index | Week of enrollment and end of the treatment at 6th weeks and 12 th weeks
Pain Assessment | Week of enrollment and end of the treatment at 6th weeks and 12 th weeks
  Visual analog scale was used to assess pain.
DASH Upper extremity Function Scale | Week of enrollment and end of the treatment at 6th weeks and 12 th weeks
Hand Grip Strenght | Week of enrollment and end of the treatment at 6th weeks and 12 th weeks
Upper Trapezius EMG Activation | Week of enrollment and end of the treatment at 6th weeks and 12 th weeks
SF-36 | Week of enrollment and end of the treatment at 6th weeks and 12 th weeks
Upper Trapezius MVC on SEMG | Week of enrollment and end of the treatment at 6th weeks and 12 th weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pervin Yeşiloğlu, Research Assisstant, Principal Investigator — Yuzuncu Yil University; Ayşe M Tat, Assoc. Prof., Study Chair — Yuzuncu Yil University; Murat Toprak, Assoc. Prof., Study Chair — Van Yüzüncü Yıl Üniversitesi Tıp Fakültesi
Locations (1):
- Dokuz Eylül üniversitesi, Izmir, Balcova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No